CLINICAL TRIAL: NCT04772950
Title: Measuring Deep and Superficial Multifidus and the Activation Pattern During Dynamic Task Correlating With Trunk Stability Ability and Functional Performance in Different Ages Asymptomatic and Unspecific Low Back Pain Adult
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202012034RINB
Record Dates: First submitted 2021-02-23; First posted 2021-02-26 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy adults
- Patients with non-specific low back pain

SUMMARY:
The first propose of the study is to understand the contraction of deep and superficial multifidus in patients with non-specific low back pain and the elderly. The second purpose of the study is to understand the relationship between the multifidus and the functional performance in patients with non-specific low back pain and the elderly. The hypothesis is that the patients with non-specific low back pain and the elderly have less ability to contract the deep multifidus then asymptomatic adults and younger adults. Besides, the multifidus is correlated to the functional performance.

ELIGIBILITY:
Inclusion Criteria:

* age 20-90
* have lumbar region discomfort in the past three months, and the discomfort is more than one day
* have diagnosis of non-specific low back pain

Exclusion Criteria:

* have received surgery of lumbar or lower extremities
* neurological symptom (eg. numbness of lower extremities)
* have no ability to stand and walking independently
* cancer
* systemic disease (eg. ankylosing spondylitis, rheumatoid arthritis, Systemic lupus erythematosus)
* pregnancy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with non-specific low back pain
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of superficial multifidus | 10 minutes
  change of superficial multifidus during contraction by using ultrasound image
Change of deep multifidus | 10 minutes
  change of deep multifidus during contraction by using ultrasound image
Disability index | 5 minutes
  use Oswestry Disability Index
Timed up and go test | 3 minutes
  Examiner will record the seconds the subjects spend in the test including standing up, walking, turn around and sit down.
Sit to stand test | 3 minutes
  Subjects will repeat 5 times sit to stand and the seconds subjects spend will be recorded.
Countermovement jump test | 3 minutes
  The subjects start from an upright standing position, makes a preliminary downward movement by flexing at the knees and hips, then immediately extends the knees and hips again to jump vertically up off the ground. The distance which the subjects jump for will be recorded.
Sahrmann five-level core stability test | 5 minutes
  Examiner will use stabilizer pressure biofeedback unit to detect whether there is lumbar motion during different levels of lower extremities movement.
Rotatory stability test | 3 minutes
  Rotatory stability test is one of the test from functional movement screen. Subjects will start in quadruped position and move the extremities to maintain the spine in neutral position.

CONTACTS AND LOCATIONS:
Locations (1):
- Shing-Tian, Chiang, Taipei, Taiwan